CLINICAL TRIAL: NCT01018186
Title: A Randomized, Double-Blind, Double Dummy, Active Comparator, Parallel Group, Multicenter Study to Evaluate the Safety of Once-Daily Fluticasone Furoate/GW642444 Inhalation Powder for 52 Weeks in Adolescent and Adult Subjects With Asthma
Brief Title: Fluticasone Furoate/GW642444 Inhalation Powder Long-Term Safety Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106839
Record Dates: First submitted 2009-11-05; First posted 2009-11-23 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone furoate/GW642444 (Experimental)
  Interventions: Drug: Fluticasone Furoate/GW642444
- Fluticasone propionate (Active Comparator)
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Fluticasone Furoate/GW642444 — Combination inhaled corticosteroid and long-acting beta2-agonist
  Arms: Fluticasone furoate/GW642444
Drug: Fluticasone propionate — Inhaled corticosteroid
  Arms: Fluticasone propionate

SUMMARY:
The purpose of this study is to evaluate the long-term safety of fluticasone furoate/GW642444

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Reversibility FEV1 of twelve percent or greater and two hundred milliliters and greater approximately ten to forty minutes following two to four inhalations of albuterol
* FEV1 greater than or equal to fifty percent of predicted
* Currently using moderate to high dose inhaled corticosteroid therapy

Exclusion Criteria:

* History of life threatening asthma
* Respiratory infection or oral candidiasis
* Asthma exacerbation
* Uncontrolled disease or clinical abnormality
* Allergies
* Taking another investigational medication or prohibited medication

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2009-10-19; Primary Completion 2011-05-01 (Actual); Study Completion 2011-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- United States (18):
  - GSK Investigational Site, Oxford, Alabama
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Greenfield, Wisconsin
- Germany (10):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Bad Woerrishofen, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Radebeul, Saxony
  - GSK Investigational Site, Reinfeld, Schleswig-Holstein
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
- Ukraine (4):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Simferopol

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Busse WW, O'Byrne PM, Bleecker ER, Lotvall J, Woodcock A, Andersen L, Hicks W, Crawford J, Jacques L, Apoux L, Bateman ED. Safety and tolerability of the novel inhaled corticosteroid fluticasone furoate in combination with the beta2 agonist vilanterol administered once daily for 52 weeks in patients >=12 years old with asthma: a randomised trial. Thorax. 2013 Jun;68(6):513-20. doi: 10.1136/thoraxjnl-2012-202606. Epub 2013 Feb 25. PMID 23440247
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 106839 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106839 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106839 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106839 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106839 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106839 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106839 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 2:2:1 ratio to Fluticasone Furoate/GW642444 Inhalation Powder (two strengths: 200/25 micrograms (µg) once daily and 100/25 µg once daily) and fluticasone propionate 500 µg twice daily, respectively.
Pre-assignment Details: Participants meeting all inclusion criteria and none of the exclusion criteria during the screening visit entered a 2-week Run-in Period for completion of Baseline safety evaluations and to obtain Baseline measures of asthma status. At Visit 2, participants were randomized to a 52-week Double-blind Treatment Period.
Groups:
- Current Asthma Therapy at a Fixed Dose: Participants were instructed to continue using an approved fixed dose of an inhaled corticosteroid (ICS) with or without an additional controller medication (i.e., long-acting beta-agonist, leukotriene modifier, etc.) for 2 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Run-in Period.
- FF/VI 100/25 µg OD: Participants received Fluticasone Furoate (FF)/Vilanterol (VI) 100/25 micrograms (µg) inhalation powder once daily (OD) in the evening via the Dry Powder Inhaler (DPI), plus a placebo via DISKUS/ACCUHALER twice daily (BID), for 52 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FF/VI 200/25 µg OD: Participants received FF/VI 200/25 µg inhalation powder OD in the evening via the DPI, plus a placebo via DISKUS/ACCUHALER BID, for 52 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FP 500 µg BID: Participants received Fluticasone Propionate (FP) 500 µg BID via DISKUS/ACCUHALER, plus a placebo via the DPI OD in the evening, for 52 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
Period: 2-week Run-in Period
Arm/Group | Current Asthma Therapy at a Fixed Dose | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Started | 617 | 0 | 0 | 0
Completed | 503 | 0 | 0 | 0
Not Completed | 114 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0 | 0
Not completed — Did Not Meet Continuation Criteria | 97 | 0 | 0 | 0
Period: 52-week Double-blind Treatment Period
Arm/Group | Current Asthma Therapy at a Fixed Dose | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Started | 0 | 201 | 202 | 100
Completed | 0 | 161 | 161 | 71
Not Completed | 0 | 40 | 41 | 29
Not completed — Adverse Event | 0 | 5 | 3 | 6
Not completed — Lack of Efficacy | 0 | 1 | 4 | 1
Not completed — Protocol Violation | 0 | 8 | 8 | 2
Not completed — Protocol-defined Stopping Criteria | 0 | 14 | 16 | 4
Not completed — Lost to Follow-up | 0 | 1 | 3 | 4
Not completed — Physician Decision | 0 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 10 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID | Total
Number analyzed (Participants) | 201 | 202 | 100 | 503
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.7 (15.85) | 38.5 (15.64) | 38.6 (15.97) | 39.0 (15.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 124 | 62 | 316
  Male | 71 | 78 | 38 | 187
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 15 | 17 | 6 | 38
  Asian - East Asian Heritage | 0 | 0 | 1 | 1
  Asian - South East Asian Heritage | 50 | 51 | 24 | 125
  Asian - Mixed Race | 0 | 0 | 1 | 1
  White - Arabic/North African Heritage | 4 | 1 | 0 | 5
  White - White/Caucasian/European Heritage | 129 | 132 | 68 | 329
  White - Mixed Race | 2 | 1 | 0 | 3
  Mixed Race | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the start of study medication until Visit 11 (Week 52)/Early Withdrawal
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
participants
  Any AE | 139 | 134 | 73
  Any SAE | 3 | 1 | 7

2. Primary Outcome: Number of Participants With Severe Asthma Exacerbations During the Treatment Period
Description: A severe asthma exacerbation is defined as the deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids. Courses of corticosteroids separated by 1 week or more were treated as separate severe exacerbations.
Time Frame: From the start of study medication until Visit 11 (Week 52)/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Groups:
- FF/VI 100/25 µg OD: Participants received FF/VI 100/25 µg inhalation powder OD in the evening via the DPI, plus a placebo via DISKUS/ACCUHALER BID, for 52 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FP 500 µg BID: Participants received FP 500 µg BID via DISKUS/ACCUHALER, plus a placebo via the DPI OD in the evening, for 52 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
participants | 3 | 6 | 3

3. Primary Outcome: Change From Baseline in Albumin and Total Protein at Week 12, Week 28, and Week 52/Early Withdrawal
Description: Blood samples were collected for the measurement of albumin and total protein values at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the most recent recorded value at Screening or prior to Day 1. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Grams per liter (G/L)
  Albumin, Week 12, n=172, 182, 87 | 0.1 (2.69) | 0.2 (2.87) | -0.5 (2.64)
  Albumin, Week 28, n=180, 176, 79 | -0.2 (2.68) | -0.3 (2.79) | -0.4 (2.76)
  Albumin, Week 52, n=157, 159, 67 | -0.1 (2.81) | -0.8 (2.72) | -0.5 (2.54)
  Total Protein, Week 12, n=172, 182, 87 | -0.6 (4.13) | -0.1 (4.50) | -0.6 (3.96)
  Total Protein, Week 28, n=180, 176, 79 | -1.1 (3.90) | -1.0 (4.47) | -0.5 (4.33)
  Total Protein, Week 52, n=157, 159, 67 | -0.7 (4.53) | -1.4 (4.60) | -1.0 (4.38)

4. Primary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase (CK), and Gamma Glutamyltransferase (GGT) at Week 12, Week 28, and Week 52/Early Withdrawal
Description: Blood samples were collected for the measurement of ALP, ALT, AST, CK, and GGT values at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the most recent recorded value at Screening or prior to Day 1. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
International units per liter (IU/L)
  ALP, Week 12, n=158, 165, 84 | -3.0 (18.76) | -2.6 (29.65) | -4.7 (24.47)
  ALP, Week 28, n=180, 176, 79 | -1.0 (32.68) | -5.8 (30.56) | -5.7 (24.33)
  ALP, Week 52, n=157, 157, 67 | -4.0 (30.67) | -7.2 (34.65) | -9.3 (27.54)
  ALT, Week 12, n=172, 182, 87 | -1.0 (10.43) | -0.2 (13.51) | -0.3 (12.03)
  ALT, Week 28, n=180, 176, 79 | -1.6 (10.08) | -0.1 (10.59) | 0.4 (11.96)
  ALT, Week 52, n=157, 159, 67 | -1.8 (12.40) | -1.3 (11.13) | -0.1 (9.78)
  AST, Week 12, n=171, 181, 87 | -0.9 (8.07) | -0.3 (12.05) | 0.3 (8.69)
  AST, Week 28, n=179, 176, 79 | -1.4 (8.42) | -0.9 (11.60) | 1.3 (10.65)
  AST, Week 52, n=156, 158, 67 | -1.8 (8.78) | -1.9 (11.21) | -0.2 (9.22)
  GGT, Week 12, n=172, 182, 87 | 0.9 (12.90) | -0.1 (18.23) | -1.7 (12.12)
  GGT, Week 28, n=180, 176, 79 | 3.3 (33.79) | -0.6 (17.63) | -0.2 (11.85)
  GGT, Week 52, n=157, 159, 67 | 2.7 (40.34) | -2.7 (15.99) | -0.5 (13.30)
  Creatinine Kinase, Week 12, n=172, 181, 87 | 10.8 (92.06) | -11.5 (254.71) | -18.3 (223.59)
  Creatinine Kinase, Week 28, n=180, 176, 79 | 2.0 (68.72) | -9.9 (247.61) | 15.3 (441.68)
  Creatinine Kinase, Week 52, n=157, 159, 67 | -0.7 (69.12) | -16.8 (266.48) | -27.7 (274.14)

5. Primary Outcome: Change From Baseline in Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, and Creatinine at Week 12, Week 28, and Week 52/Early Withdrawal
Description: Blood samples were collected for the measurement of direct bilirubin, indirect bilirubin, total bilirubin, and creatinine values at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the most recent recorded value at Screening or prior to Day 1. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Micromoles per liter (µmol/L)
  Direct bilirubin, Week 12, n=172, 182, 87 | -0.3 (0.99) | -0.3 (0.98) | -0.2 (0.93)
  Direct bilirubin, Week 28, n=180, 176, 79 | -0.3 (0.97) | -0.2 (1.01) | -0.1 (0.94)
  Direct bilirubin, Week 52, n=157, 159, 67 | -0.4 (0.99) | -0.4 (1.00) | -0.2 (0.90)
  Indirect bilirubin, Week 12, n=172, 182, 87 | -1.4 (3.11) | -0.8 (2.86) | -0.6 (3.04)
  Indirect bilirubin, Week 28, n=180, 175, 79 | -1.3 (3.09) | -0.9 (2.87) | -0.4 (3.14)
  Indirect bilirubin, Week 52, n=157, 159, 67 | -2.0 (3.08) | -1.6 (2.51) | -0.8 (2.68)
  Total Bilirubin, Week 12, n=172, 182, 87 | -1.7 (3.62) | -1.1 (3.46) | -0.8 (3.44)
  Total Bilirubin, Week 28, n=180, 175, 79 | -1.6 (3.61) | -1.2 (3.55) | -0.5 (3.46)
  Total Bilirubin, Week 52, n=157, 159, 67 | -2.4 (3.58) | -2.0 (2.93) | -1.0 (3.14)
  Creatinine, Week 12, n=172, 181, 87 | 3.00 (10.214) | 3.18 (7.983) | 3.99 (8.056)
  Creatinine, Week 28, n=180, 176, 79 | 7.03 (19.264) | 5.10 (10.316) | 17.43 (92.175)
  Creatinine, Week 52, n=157, 159, 67 | 2.74 (9.450) | 3.14 (11.310) | 3.32 (9.982)

6. Primary Outcome: Change From Baseline in Chloride, Carbon Dioxide Content/Bicarbonate, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) at Week 12, Week 28, and Week 52/Early Withdrawal
Description: Blood samples were collected for the measurement of chloride, carbon dioxide (CO2) content/bicarbonate, glucose, potassium, sodium, and urea/BUN values at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the most recent recorded value at Screening or prior to Day 1. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Millimoles per liter (mmol/L)
  Chloride, Week 12, n=172, 182, 87 | -0.7 (3.43) | -0.4 (3.50) | 0.1 (2.28)
  Chloride, Week 28, n=180, 176, 79 | -0.1 (2.50) | 0.2 (2.73) | -0.1 (2.54)
  Chloride, Week 52, n=157, 159, 67 | -0.5 (2.51) | 0.0 (2.67) | -0.3 (2.31)
  CO2 content/bicarbonate, Week 12, n=171, 181, 87 | -0.7 (3.13) | -0.8 (2.91) | -0.2 (2.72)
  CO2 content/bicarbonate, Week 28, n=179, 176, 79 | 0.3 (2.90) | 0.1 (2.61) | 0.9 (2.60)
  CO2 content/bicarbonate, Week 52, n=156, 158, 67 | -0.1 (2.53) | 0.1 (2.51) | 0.5 (2.55)
  Glucose, Week 12, n=172, 181, 87 | 0.33 (1.873) | 0.17 (2.085) | 0.10 (1.233)
  Glucose, Week 28, n=180, 175, 79 | 0.21 (1.547) | 0.16 (1.556) | 0.02 (1.442)
  Glucose, Week 52, n=157, 159, 67 | 0.45 (1.839) | 0.11 (1.426) | -0.20 (1.191)
  Potassium, Week 12, n=157, 165, 84 | -0.09 (0.572) | 0.00 (0.721) | -0.03 (0.606)
  Potassium, Week 28, n=179, 176, 79 | -0.12 (0.467) | -0.15 (0.449) | 0.02 (0.617)
  Potassium, Week 52, n=156, 156, 67 | -0.18 (0.461) | -0.12 (0.535) | -0.10 (0.446)
  Sodium, Week 12, n=172, 182, 87 | -0.1 (2.47) | 0.2 (2.61) | -0.0 (2.24)
  Sodium, Week 28, n=180, 176, 79 | 0.0 (2.46) | 0.2 (2.65) | 0.3 (2.74)
  Sodium, Week 52, n=157, 159, 67 | -0.2 (2.57) | 0.1 (2.52) | 0.0 (2.80)
  Urea/BUN, Week 12, n=172, 182, 87 | 0.24 (1.299) | 0.36 (1.237) | 0.02 (1.757)
  Urea/BUN, Week 28, n=180, 176, 79 | 0.16 (1.460) | 0.14 (1.124) | 0.41 (2.676)
  Urea/BUN, Week 52, n=157, 159, 67 | 0.15 (1.244) | 0.13 (1.479) | -0.04 (1.900)

7. Primary Outcome: Change From Baseline in the Percentage of Basophils, Eosinophils, Hematocrit, Lymphocytes, Monocytes, and Segmented Neutrophils in the Blood at Week 12, Week 28, and Week 52/Early Withdrawal
Description: Blood samples were collected for the measurement of the percentage of basophils, eosinophils, hematocrit, lymphocytes, monocytes, and segmented neutrophils in the blood at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the most recent recorded value at Screening or prior to Day 1. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 101
Percentage
  Basophils, Week 12, n=171, 170, 86 | -0.01 (0.330) | -0.06 (0.331) | -0.08 (0.320)
  Basophils, Week 28, n=169, 169, 77 | -0.01 (0.319) | 0.00 (0.338) | -0.06 (0.310)
  Basophils, Week 52, n=155, 155, 71 | 0.02 (0.314) | -0.03 (0.279) | -0.07 (0.319)
  Eosinophils, Week 12, n=171, 170, 86 | -0.35 (4.048) | -0.88 (3.825) | -1.23 (3.391)
  Eosinophils, Week 28, n=169, 169, 77 | -0.97 (3.991) | -1.34 (3.774) | -1.63 (3.574)
  Eosinophils, Week 52, n=155, 155, 71 | -0.84 (4.096) | -0.90 (3.946) | -1.19 (3.611)
  Lymphocytes, Week 12, n=171, 170, 86 | -0.57 (9.280) | -0.91 (8.414) | -1.72 (8.449)
  Lymphocytes, Week 28, n=169, 169, 77 | -1.11 (8.816) | -1.31 (10.200) | -1.66 (11.054)
  Lymphocytes, Week 52, n=155, 155, 71 | 1.34 (9.389) | -0.03 (10.137) | -0.97 (8.532)
  Monocytes, Week 12, n=171, 170, 86 | -0.60 (2.692) | -0.47 (2.500) | -0.86 (3.147)
  Monocytes, Week 28, n=169, 169, 77 | -0.66 (2.594) | -0.53 (2.706) | -0.84 (3.063)
  Monocytes, Week 52, n=155, 155, 71 | -0.19 (2.439) | 0.31 (2.598) | -0.30 (2.337)
  Segmented neutrophils, Week 12, n=171, 170, 86 | 1.54 (10.883) | 2.32 (9.635) | 3.89 (11.397)
  Segmented neutrophils, Week 28, n=169, 169, 77 | 2.71 (10.221) | 3.18 (12.008) | 4.19 (13.745)
  Segmented neutrophils, Week 52, n=155, 155, 71 | -0.33 (10.687) | 0.66 (11.768) | 2.54 (10.112)

8. Primary Outcome: Change From Baseline in Eosinophil Count, Total Absolute Neutrophil Count (ANC), Platelet Count, and White Blood Cell (WBC) Count at Week 12, Week 28, and Week 52/Early Withdrawal
Description: Blood samples were collected to determine the eosinophil count, total ANC, platelet count, and WBC count at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the most recent recorded value at Screening or prior to Day 1. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
10^9 cells per liter (GI/L)
  Eosinophil count, Week 12, n=171, 170, 86 | -0.010 (0.3226) | -0.057 (0.3841) | -0.073 (0.2220)
  Eosinophil count, Week 28, n=169, 169, 77 | -0.039 (0.3310) | -0.083 (0.3698) | -0.083 (0.2363)
  Eosinophil count, Week 52, n=155, 155, 71 | -0.023 (0.3273) | -0.037 (0.3171) | -0.044 (0.2539)
  Total ANC, Week 12, n=171, 170, 86 | 0.392 (1.6161) | 0.469 (1.6904) | 0.493 (1.7488)
  Total ANC, Week 28, n=169, 169, 77 | 0.632 (1.5922) | 0.679 (2.0157) | 0.750 (2.0130)
  Total ANC, Week 52, n=136, 136, 60 | 0.524 (1.4589) | 0.612 (1.9100) | 0.748 (1.7946)
  Platelet Count, Week 12, n=167, 159, 78 | -1.3 (39.44) | 1.5 (68.10) | 1.5 (43.26)
  Platelet Count, Week 28, n=164, 165, 74 | 1.0 (44.49) | 3.5 (35.06) | 12.4 (43.59)
  Platelet Count, Week 52, n=147, 151, 68 | 1.8 (43.80) | 4.6 (38.49) | 16.4 (50.99)
  WBC Count, Week 12, n=173, 170, 86 | 0.51 (1.744) | 0.50 (2.007) | 0.39 (1.906)
  WBC Count, Week 28, n=170, 169, 77 | 0.74 (1.758) | 0.74 (2.103) | 0.79 (2.028)
  WBC Count, Week 52, n=156, 156, 71 | 0.91 (1.639) | 0.83 (2.046) | 1.01 (1.909)

9. Primary Outcome: Change From Baseline in Hematocrit at Week 12, Week 28, and Week 52/Early Withdrawal
Description: Blood samples were collected for the measurement of hematocrit values at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the most recent recorded value at Screening or prior to Day 1. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Proportion of 1.0
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Proportion of 1.0
  Week 12, n=176, 172, 86 | -0.0073 (0.02307) | -0.0013 (0.02654) | -0.0025 (0.02318)
  Week 28, n=172, 170, 77 | -0.0017 (0.02213) | -0.0005 (0.02464) | -0.0028 (0.02168)
  Week 52, n=157, 159, 72 | -0.0027 (0.02906) | -0.0021 (0.02467) | -0.0045 (0.02495)

10. Primary Outcome: Change From Baseline in Hemoglobin at Week 12, Week 28, and Week 52/Early Withdrawal
Description: Blood samples were collected for the measurement of hemoglobin values at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the most recent recorded value at Screening or prior to Day 1. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Groups:
- FF/VI 200/25 µg OD: Participants received FF/VI 200/25 µg inhalation powder OD in the evening via the DPI, plus a placebo via DISKUS/ACCUHALER BID, for 52 weeks. Participnts were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FP 500 µg BID: Participants received FP 500 µg BID via DISKUS/ACCUHALER, plus a placebo via the DPI OD in the evening, for 52 weeks. Participants were provided albutero/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Grams per liter (g/L)
  Week 12, n=176, 172, 86 | -3.4 (7.48) | -1.8 (8.25) | -2.0 (7.67)
  Week 28, n=172, 170, 77 | -2.1 (7.64) | -2.2 (8.11) | -2.4 (7.72)
  Week 52, n=157, 159, 72 | -2.6 (10.26) | -2.9 (7.47) | -3.0 (8.77)

11. Primary Outcome: Number of Participants With the Indicated Shift From Baseline to High, Normal or no Change, and Low Post-Baseline Values for Urinary Cortisol Excretion
Description: A 24-hour urine sample was collected for the measurement of 24-hour urinary cortisol excretion (UCE) at the following scheduled time points: Baseline, Week 12, Week 28, and Week 52/Early Withdrawal. Any visit post-baseline (AVPB) value was derived using laboratory assessments performed at scheduled, unscheduled, and Early Withdrawal visits. Participants who had a shift from Baseline in their post-Baseline UCE values relative to the normal range, are presented in the "To high and To low" categories. Participants whose post-Baseline UCE values were unchanged (e.g., High to High) or whose value became normal, are presented in the "To normal or no change" category. The normal range for UCE is defined as: 11 to 138 nanomoles per 24 hours (nmol/24 hr) for participants >=18 years of age, 8.3 to 151.7 nmol/24 hr for participants 14 to 17 years of age, and 2.8 to 124.2 nmol/24 hr for participants 12 and 13 years of age.
Time Frame: Baseline; Week 12, Week 28, and Week 52/Early Withdrawal
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
participants
  Week 12: To high, n=139, 140, 78 | 6 [4.5 to 160.6] | 7 [5.9 to 491.8] | 2 [5.3 to 780.5]
  Week 12: To normal or no change, n=139, 140, 78 | 131 [5.7 to 547.4] | 128 [6.1 to 482.5] | 67 [3.8 to 667.5]
  Week 12: To low, n=139, 140, 78 | 2 [4.0 to 602.3] | 5 [10.4 to 549.6] | 9 [3.4 to 396.4]
  Week 28: To high, n=135, 131, 59 | 8 | 8 | 3
  Week 28: To normal or no change, n=135, 131, 59 | 123 | 120 | 47
  Week 28: To low, n=135, 131, 59 | 4 | 3 | 9
  Week 52: To high, n=134, 140, 65 | 10 | 7 | 4
  Week 52: To normal or no change , n=134, 140, 65 | 119 | 131 | 57
  Week 52: To low, n=134, 140, 65 | 5 | 2 | 4
  AVBP: To high, n=156, 156, 83 | 25 | 21 | 8
  AVBP: To normal or no change, n=156, 156, 83 | 119 | 126 | 58
  AVBP: To low, n=156, 156, 83 | 12 | 9 | 17
Statistical Analysis 1: Comparison: FF/VI 100/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; Ratio = 1.67, 95% CI 2-sided [1.34 to 2.08] — Ratio of FF/VI 100/25 OD versus FP 500 BD to Baseline of 24-Hour Urinary Cortisol Excretion at Week 12
Statistical Analysis 2: Comparison: FF/VI 100/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; Ratio = 1.65, 95% CI 2-sided [1.29 to 2.13] — Ratio of FF/VI 100/25 OD versus FP 500 BD to Baseline of 24-Hour Urinary Cortisol Excretion at Week 28
Statistical Analysis 3: Comparison: FF/VI 100/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; Ratio = 1.05, 95% CI 2-sided [0.83 to 1.33] — Ratio of FF/VI 100/25 OD versus FP 500 BD to Baseline of 24-Hour Urinary Cortisol Excretion at Week 52
Statistical Analysis 4: Comparison: FF/VI 200/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; Ratio = 1.52, 95% CI 2-sided [1.22 to 1.89] — Ratio of FF/VI 200/25 OD versus FP 500 BD to Baseline of 24-Hour Urinary Cortisol Excretion at Week 12
Statistical Analysis 5: Comparison: FF/VI 200/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; Ratio = 1.43, 95% CI 2-sided [1.11 to 1.84] — Ratio of FF/VI 200/25 OD versus FP 500 BD to Baseline of 24-Hour Urinary Cortisol Excretion at Week 28
Statistical Analysis 6: Comparison: FF/VI 200/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; Ratio = 1.09, 95% CI 2-sided [0.87 to 1.38] — Ratio of FF/VI 200/25 OD versus FP 500 BD to Baseline of 24-Hour Urinary Cortisol Excretion at Week 52

12. Primary Outcome: Ratio of 24-hour Urinary Cortisol Excretion at Week 12 to Baseline
Description: A 24-hour urine sample was collected, and the least square geometric mean (LSGM) for 24-hour urinary cortisol excretion (UCE) was calculated at Baseline and at Week 12. The ratio of the Week 12 LSGM to the Baseline LSGM was calculated as the value at Week 12 divided by the value at Baseline. Analysis was performed using analysis of covariance (ANCOVA) with covariates of region, sex, age, treatment, and the log of the Baseline values.
Time Frame: Baseline and Week 12
Population: Urinary cortisol (UC) Population: participants in the ITT Population whose urine samples did not have confounding factors that affected the interpretation of results. These participants were determined prior to breaking the blind. Only those participants available at the specified time point were analyzed.
Measure: Number; unit: Ratio of LSGM of UCE to Baseline
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 129 | 129 | 71
Ratio of LSGM of UCE to Baseline | 1.03 | 0.93 | 0.61
Statistical Analysis 1: Comparison: FF/VI 100/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of LSGM to Baseline = 1.67, 95% CI 2-sided [1.34 to 2.08]
Statistical Analysis 2: Comparison: FF/VI 200/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of LSGM to Baseline = 1.52, 95% CI 2-sided [1.22 to 1.89]

13. Primary Outcome: Ratio of 24-hour Urinary Cortisol Excretion at Week 28 to Baseline
Description: A 24-hour urine sample was collected, and the LSGM for 24-hour UCE was calculated at Baseline and at Week 28. The ratio of the Week 28 LSGM to the Baseline LSGM was calculated as the value at Week 28 divided by the value at Baseline. Analysis was performed using ANCOVA with covariates of region, sex, age, treatment, and the log of the Baseline values.
Time Frame: Baseline and Week 28
Population: UC Population. Only those participants available at the specified time point were analyzed.
Measure: Number; unit: Ratio of LSGM of UCE to Baseline
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 128 | 121 | 56
Ratio of LSGM of UCE to Baseline | 1.05 | 0.91 | 0.64
Statistical Analysis 1: Comparison: FF/VI 100/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of LSGM to Baseline = 1.65, 95% CI 2-sided [1.29 to 2.13]
Statistical Analysis 2: Comparison: FF/VI 200/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; p = 0.006, ANCOVA; Ratio of LSGM to Baseline = 1.43, 95% CI 2-sided [1.11 to 1.84]

14. Primary Outcome: Ratio of 24-hour Urinary Cortisol Excretion at Week 52 to Baseline
Description: A 24-hour urine sample was collected, and the LSGM for 24-hour UCE was calculated at Baseline and at Week 52. The ratio of the Week 52 LSGM to the Baseline LSGM was calculated as the value at Week 52 divided by the value at Baseline. Analysis was performed using ANCOVA with covariates of region, sex, age, treatment, and the log of the Baseline values.
Time Frame: Baseline and Week 52
Population: UC Population. Only those participants available at the specified time point were analyzed.
Measure: Number; unit: Ratio of LSGM of UCE to Baseline
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 125 | 127 | 60
Ratio of LSGM of UCE to Baseline | 1.00 | 1.04 | 0.95
Statistical Analysis 1: Comparison: FF/VI 100/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; p = 0.674, ANCOVA; Ratio of LSGM to Baseline = 1.05, 95% CI 2-sided [0.83 to 1.33]
Statistical Analysis 2: Comparison: FF/VI 200/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; p = 0.444, ANCOVA; Ratio of LSGM to Baseline = 1.09, 95% CI 2-sided [0.87 to 1.38]

15. Primary Outcome: Number of Participants With Evidence of Oral Candidiasis at Any Time Post-Baseline
Description: A detailed oropharyngeal examination was done at all clinic visits for visual/clinical evidence of oral candidiasis over the entire Treatment Period (worst case any time post-Baseline). For participants with visual/clinical evidence of candidiasis during the Treatment Phase of the study, a culture swab was taken and analyzed for infection.
Time Frame: From Baseline until Visit 11/Early Withdrawal (52 weeks)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 199 | 200 | 100
participants
  Evidence of oral candidiasis | 15 | 14 | 5
  Positive culture swab | 13 | 11 | 3
  Negative culture swab | 1 | 2 | 2
  No swab result available | 1 | 1 | 0

16. Primary Outcome: Maximum Change From Baseline in Systolic Blood Pressure (SBP) and Minimum Change From Baseline in Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured at the following scheduled time points: Screening, Day 1, Week 2, Week 4, Week 8, Week 12, Week 20, Week 28, Week 36, Week 44, and Week 52/Early Withdrawal. Baseline is defined as the Visit 1 (screening) value. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline. Maximum and minimum change from Baseline for any post-Baseline visit was derived using all scheduled, unscheduled, and Early Withdrawal visits.
Time Frame: From Baseline until Visit 11/Early Withdrawal (52 weeks)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Millimeters of mercury (mmHg)
  Maximum post-Baseline change in SBP | 10.2 (11.05) | 10.0 (10.17) | 11.3 (11.09)
  Minimum post-Baseline change in DBP | -8.9 (7.70) | -9.0 (8.44) | -8.0 (7.76)

17. Primary Outcome: Maximum Change From Baseline in Pulse Rate
Description: Pulse rate was measured at the following scheduled time points: Screening, Day 1, Week 2, Week 4, Week 8, Week 12, Week 20,Week 28, Week 36, Week 44, and Week 52/Early Withdrawal. Baseline is defined as the Visit 1 (screening) value. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline. Maximum change from Baseline for any post-Baseline visit was derived using all scheduled, unscheduled, and Early Withdrawal visits.
Time Frame: From Baseline until Visit 11/Early Withdrawal (52 weeks)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Beats per minute | 10.5 (9.30) | 10.0 (10.05) | 7.5 (8.29)

18. Primary Outcome: Number of Participants With the Indicated Change From Baseline in Lens Opacities Classification System, Version III (LOCS III) Posterior Subcapsular Opacity (P) at Week 28 and Week 52
Description: P is defined as the opacification at the back of the lens adjacent to the capsule (or bag) in which the lens sits. An event of P is defined as an increase of >=0.3 from Baseline in LOCS III grade for P in either eye at any time post-Baseline. Per LOC III, P ranges from 0.1 (clear or colorless) to 5.9 (very opaque). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 28, and Week 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
participants
  Left eye, <0.3, Week 28, n=179, 177, 80 | 174 | 175 | 79
  Left eye, >=0.3 and <0.5, Week 28, n=179, 177, 80 | 5 | 2 | 1
  Left eye, >=0.5, Week 28, n=179, 177, 80 | 0 | 0 | 0
  Right eye, <0.3, Week 28, n=179, 177, 80 | 175 | 175 | 80
  Right eye, >=0.3 and <0.5, Week 28, n=179, 177, 80 | 4 | 2 | 0
  Right eye, >=0.5, Week 28, n=179, 177, 80 | 0 | 0 | 0
  Left eye, <0.3, Week 52, n=167, 166, 72 | 163 | 164 | 72
  Left eye, >=0.3 and <0.5, Week 52, n=167, 166, 72 | 2 | 1 | 0
  Left eye, >=0.5, Week 52, n=167, 166, 72 | 2 | 1 | 0
  Right eye, <0.3, Week 52, n=167, 166, 72 | 163 | 164 | 72
  Right eye, >=0.3 and <0.5, Week 52, n=167, 166, 72 | 3 | 1 | 0
  Right eye, >=0.5, Week 52, n=167, 166, 72 | 1 | 1 | 0

19. Primary Outcome: Number of Participants With the Indicated Change From Baseline in Intraocular Pressure (IOP) at Week 28 and Week 52
Description: Intraocular pressure (IOP) is the fluid pressure inside the eye. IOP was measured twice for each eye at Baseline, Week 28, and Week 52 using Goldmann Applanation tonometry. The second IOP reading was used for analysis. The number of participants with a change from Baseline in IOP of <0 mmHg, >=0 to <4 mmHg, >=4 to <7 mmHg, >=7 to <11 mmHg, and >=11 mmHg are presented. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 28 and Week 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
participants
  Left eye, <0 mmHg, Week 28, n=179, 177, 80 | 71 | 78 | 32
  Left eye, >=0 to <4 mmHg, Week 28, n=179, 177, 80 | 101 | 92 | 46
  Left eye, >=4 to <7 mmHg, Week 28, n=179, 177, 80 | 7 | 6 | 2
  Left eye, >=7 to <11 mmHg, Week 28, n=179, 177, 80 | 0 | 1 | 0
  Left eye, >=11 mmHg, Week 28, n=179, 177, 80 | 0 | 0 | 0
  Right eye, <0 mmHg, Week 28, n=179, 177, 80 | 73 | 61 | 38
  Right eye, >=0 to <4 mmHg, Week 28, n=179, 177, 80 | 101 | 110 | 38
  Right eye, >=4 to <7 mmHg, Week 28, n=179, 177, 80 | 5 | 5 | 4
  Right eye, >=7 to <11 mmHg,Week 28, n=179, 177, 80 | 0 | 1 | 0
  Right eye, >=11 mmHg, Week 28, n=179, 177, 80 | 0 | 0 | 0
  Left eye, <0 mmHg, Week 52, n=167, 166, 72 | 66 | 69 | 33
  Left eye, >=0 to <4 mmHg, Week 52, n=167, 166, 72 | 88 | 83 | 36
  Left eye, >=4 to <7 mmHg, Week 52, n=167, 166, 72 | 11 | 14 | 3
  Left eye, >=7 to <11 mmHg, Week 52, n=167, 166, 72 | 2 | 0 | 0
  Left eye, >=11 mmHg, Week 52, n=167, 166, 72 | 0 | 0 | 0
  Right eye, <0 mmHg, Week 52, n=167, 166, 72 | 63 | 61 | 32
  Right eye, >=0 to <4 mmHg, Week 52, n=167, 166, 72 | 94 | 93 | 40
  Right eye, >=4 to <7 mmHg, Week 52, n=167, 166, 72 | 10 | 12 | 0
  Right eye, >=7 to <11 mmHg, Week 52, n=167,166, 72 | 0 | 0 | 0
  Right eye, >=11 mmHg, Week 52, n=167, 166, 72 | 0 | 0 | 0

20. Primary Outcome: Change From Baseline in Horizontal Cup-to-disc Ratio at Week 28 and Week 52
Description: Funduscopic examination was performed at Baseline, Week 28, and Week 52 to measure the horizontal cup-to-disc ratio of both eyes. The horizontal cup-to-disc ratio is the ratio of the horizontal diameter of the physiological cup to that of the horizontal diameter of the optic disc. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 28 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
ratio
  Left eye, Week 28, n=179, 177, 80 | 0.5 (4.79) | -0.2 (5.11) | 0.5 (4.87)
  Right eye, Week 28, n=179, 177, 80 | 0.2 (4.17) | -0.2 (6.49) | 0.5 (5.10)
  Left eye, Week 52, n=167, 166, 72 | 0.4 (5.86) | 0.2 (4.89) | 0.3 (4.77)
  Right eye, Week 52, n=167, 166, 72 | 0.1 (4.63) | 0.2 (5.57) | 0.0 (5.26)

21. Primary Outcome: Number of Participants With the Indicated Change From Baseline in Lens Opacities Classification System, Version III (LOCS III) Cortical Opacity (C) at Week 28 and Week 52
Description: C is defined as the opacification of the cortex (outer layer) of the lens. Per LOC III, C ranges from 0.1 (clear or colorless) to 5.9 (very opaque). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 28 and Week 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
participants
  Left eye, <0.3, Week 28, n=179, 177, 80 | 167 | 166 | 75
  Left eye, >=0.3 and <0.5, Week 28, n=179, 177, 80 | 6 | 5 | 4
  Left eye, >=0.5, Week 28, n=179, 177, 80 | 6 | 6 | 1
  Right eye, <0.3, Week 28, n=179, 177, 80 | 169 | 172 | 75
  Right eye, >=0.3 and <0.5, Week 28, n=179, 177, 80 | 5 | 1 | 4
  Right eye, >=0.5, Week 28, n=179, 177, 80 | 5 | 4 | 1
  Left eye, <0.3, Week 52, n=167, 166, 72 | 154 | 156 | 66
  Left eye, >=0.3 and <0.5, Week 52, n=167, 166, 72 | 7 | 4 | 3
  Left eye, >=0.5, Week 52, n=167, 166, 72 | 6 | 6 | 3
  Right eye, <0.3, Week 52, n=167, 166, 72 | 151 | 158 | 69
  Right eye, >=0.3 and <0.5, Week 52, n=167, 166, 72 | 11 | 2 | 2
  Right eye, >=0.5, Week 52, n=167, 166, 72 | 5 | 6 | 1

22. Primary Outcome: Change From Baseline in Lens Opacities Classification System, Version III (LOCS III) Nuclear Color (NC) at Week 28 and Week 52
Description: NC is the color of the nucleus (central layer) of the lens. Per LOC III, NC ranges from 0.1 (clear or colorless) to 6.9 (very opaque or brunescent). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 28 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Scores on a scale
  Week 28, Left eye, n=179, 177, 80 | 0.01 (0.282) | 0.00 (0.284) | -0.02 (0.299)
  Week 28, Right eye, n=179, 177, 80 | 0.01 (0.292) | 0.1 (0.292) | -0.02 (0.294)
  Week 52, Left eye, n=167, 166, 72 | 0.02 (0.281) | -0.2 (0.357) | 0.00 (0.340)
  Week 52, Right eye, n=167, 166, 72 | 0.02 (0.304) | 0.00 (0.339) | 0.01 (0.336)

23. Primary Outcome: Change From Baseline in Lens Opacities Classification System, Version III (LOCS III) Nuclear Opalescence (NO) at Week 28 and Week 52
Description: NO is the opalescence of the nucleus (central layer) of the lens. Per LOC III, NO ranges from 0.1 (clear or colorless) to 6.9 (very opaque or brunescent). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 28 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Scores on a scale
  Week 28, Left eye, n=179, 177, 80 | 0.02 (0.236) | 0.03 (0.316) | -0.02 (0.270)
  Week 28, Right eye, n=179, 177, 80 | 0.01 (0.256) | 0.03 (0.303) | -0.03 (0.272)
  Week 52, Left eye, n=167, 166, 72 | 0.01 (0.330) | 0.03 (0.303) | 0.01 (0.369)
  Week 52, Right eye, n=167, 166, 72 | 0.00 (0.351) | 0.04 (0.282) | 0.02 (0.371)

24. Primary Outcome: Change From Baseline in the Logarithm of the Minimum Angle of Resolution (LogMAR) Visual Acuity at Week 28 and Week 52
Description: Visual acuity is defined as the acuteness or clearness of vision. The minimum angle of resolution (MAR) is the angle a viewed object subtends at the eye, usually stated in degrees/minutes of arc. Visual acuity was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) charts in decimal numbers. The LogMAR scale is used to express the visual acuity in a linear scale as the logarithm to base 10 of the MAR. A lower score indicates better visual acuity; visual acuity decreases with an increasing score. Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline; Week 28 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
Scores on a scale
  Week 28, Left eye, n=179, 176, 80 | -0.008 (0.0723) | -0.010 (0.0706) | -0.004 (0.0685)
  Week 28, Right eye, n=179, 176, 80 | -0.003 (0.0739) | -0.001 (0.0699) | -0.008 (0.0584)
  Week 52, Left eye, n=167, 165, 72 | -0.011 (0.0747) | -0.012 (0.0739) | -0.007 (0.0638)
  Week 52, Right eye, n=167, 165, 72 | -0.008 (0.0928) | 0.003 (0.0755) | -0.012 (0.0776)

25. Primary Outcome: Maximum Change From Baseline in the QT Interval Using Bazett's Correction (QTcB) and QT Interval Using Fridericia's Correction (QTcF)
Description: The QT interval is an electrocardiogram (ECG) parameter that represents the electrical depolarization and repolarization of the left and right ventricles of the heart. The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the ECG. Corrected QT (QTc) is the QT interval corrected for heart rate by using Bazett's formula (QTcB) and Fridericia's formula (QTcF). 12-lead ECG measurements were perfomed at the following scheduled time points: Baseline; Week 2, Week 12, Week 28, and Week 52/Early Withdrawal. The Baseline value is defined as the value taken pre-dose at screening. The maximum post-Baseline value was derived using all scheduled, unscheduled, and Early Withdrawal ECG assessments. Maximum change from Baseline was calculated as the maximum post-Baseline value minus the value at Baseline.
Time Frame: Baseline; Week 2, Week 12, Week 28, and Week 52/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 199 | 198 | 100
Milliseconds (msec)
  QTcB | 19.0 (17.33) | 16.4 (19.49) | 13.2 (16.57)
  QTcF | 12.8 (14.51) | 11.6 (15.60) | 11.4 (12.81)

26. Primary Outcome: Mean 24 Hour Holter Heart Rate for Participants With at Least 16 Hours of Recorded Data
Description: Twenty-four hour Holter monitors were obtained using a 12-lead Holter monitor. The Holter monitor is worn by the participant for 24 hours, and the monitor continuously records the heart's rhythm while the monitor is worn. At the end of the 24 hour period, the data from the monitor are downloaded and transmitted to the centralized vendor for analysis and interpretation by a licensed cardiologist.
Time Frame: 0-24 hours at Screening, Day 1, Week 28, and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
beats per minute
  Screening, n=111, 116, 49 | 79.0 (8.23) | 79.1 (9.55) | 79.8 (8.75)
  Day 1, n=104, 113, 47 | 78.6 (7.89) | 78.7 (9.45) | 77.4 (7.66)
  Week 28, n=95, 90, 39 | 77.8 (8.90) | 77.5 (9.01) | 74.9 (8.54)
  Week 52, n=88, 82, 37 | 78.8 (8.72) | 78.0 (10.15) | 74.8 (8.62)

27. Primary Outcome: Maximum 24 Hour Holter Heart Rate for Participants With at Least 16 Hours of Recorded Data
Description: Twenty-four hour Holter monitors were obtained using a 12-lead Holter monitor. Holter monitor data were transmitted to a centralized vendor for analysis and interpretation by a licensed cardiologist.
Time Frame: 0-24 hours at Screening, Day 1, Week 28, and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 201 | 202 | 100
beats per minute
  Screening, n=111, 116, 49 | 132.6 (17.18) | 132.1 (17.85) | 133.0 (16.17)
  Day 1, n=104, 113, 47 | 131.2 (18.28) | 130.8 (19.50) | 129.2 (18.77)
  Week 28, n=95, 90, 39 | 127.5 (17.93) | 127.4 (16.62) | 123.5 (14.93)
  Week 52, n=88, 82, 37 | 126.9 (18.16) | 128.1 (16.63) | 122.8 (13.89)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until Follow-up (up to 52 weeks of treatment).
Description: SAEs and non-serious AEs were collected in the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Groups:
- FP 500 µg BD: Participants received Fluticasone Propionate (FP) 500 µg BID via DISKUS/ACCUHALER, plus a placebo via the DPI OD in the evening, for 52 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
Arm/Group | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | FP 500 µg BD
Serious Adverse Events (participants affected / at risk) | 3/201 | 1/202 | 7/100
Other Adverse Events (participants affected / at risk) | 108/201 | 105/202 | 61/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg OD (N=201) | FF/VI 200/25 µg OD (N=202) | FP 500 µg BD (N=100)
Dengue Fever (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg OD (N=201) | FF/VI 200/25 µg OD (N=202) | FP 500 µg BD (N=100)
Upper respiratory tract infection (Infections and infestations) | 34 | 30 | 18
Nasopharyngitis (Infections and infestations) | 25 | 19 | 10
Oral candidiasis (Infections and infestations) | 12 | 11 | 2
Bronchitis (Infections and infestations) | 7 | 9 | 5
Respiratory tract infection (Infections and infestations) | 6 | 5 | 7
Sinusitis (Infections and infestations) | 9 | 4 | 5
Headache (Nervous system disorders) | 39 | 35 | 23
Tension headache (Nervous system disorders) | 1 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 11 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 8 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 13 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3
Pyrexia (General disorders) | 8 | 13 | 6
Extrasystoles (Cardiac disorders) | 4 | 15 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.